CLINICAL TRIAL: NCT04289285
Title: Safety and Efficacy of IBI306 in Chinese Non-familial Hypercholesterolemia Subjects at Very High or High Cardiovascular Risk: a Randomized, Double-blind and Placebo-controlled Phase III Study
Brief Title: Safety and Efficacy of IBI306 in Chinese Subjects With Non-familial Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI306B301
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IBI306 450mg SC Q4W (Experimental)
  Interventions: Drug: IBI306 450mg SC Q4W
- Placebo SC Q4W (Placebo Comparator)
  Interventions: Drug: Placebo SC Q4W
- IBI306 600mg SC Q6W (Experimental)
  Interventions: Drug: IBI306 600mg SC Q6W
- Placebo SC Q6W (Placebo Comparator)
  Interventions: Other: Placebo SC Q6W

INTERVENTIONS:
Drug: IBI306 450mg SC Q4W — Subjects will receive IBI306 450mg every 4 weeks subcutaneously.
  Arms: IBI306 450mg SC Q4W
Drug: Placebo SC Q4W — Subjects will receive placebo every 4 weeks subcutaneously.
  Arms: Placebo SC Q4W
Drug: IBI306 600mg SC Q6W — Subjects will receive IBI306 600mg every 6 weeks subcutaneously.
  Arms: IBI306 600mg SC Q6W
Other: Placebo SC Q6W — Subjects will receive placebo every 6 weeks subcutaneously.
  Arms: Placebo SC Q6W

SUMMARY:
IBI306 is a fully human monoclonal antibody that binds proprotein convertase substilisin/kexin type 9 (PCSK-9), preventing its interaction with the low-density lipoprotein cholesterol receptor (LDL-R) and thereby restoring LDL-R recycling and low-density lipoprotein cholesterol(LDL-C) uptake. This study is being done to investigate the effects of IBI306 in Chinese people with non-familial hypercholesterolemia with very high or high cardiovascular risk. This study will see if IBI306 will reduce low density lipoprotein cholesterol (LDL-C) in Chinese people who are taking a certain type of lipid-lowering medication (statins with or without ezetimibe) and whether it causes any side effects

DETAILED DESCRIPTION:
This is a phase 3, multicenter, double-blind, randomized, placebo-controlled study of IBI306 in Chinese non-familial hypercholesterolemia Subjects with very high or high cardiovascular risk. A total of around 600 subjects who meet admission criteria will be randomized and receive one of the two dose levels of IBI306 or matching placebo: 450mg Q4W, or 600mg Q6W. The double blind period for both groups will be 48 weeks. The study will last 52 weeks

ELIGIBILITY:
Inclusion criteria:

1. Males and females ≥ 18 to ≤ 75 years of age
2. Diagnosis of hypercholesterolemia
3. LDL cholesterol ≥ 70 mg/dl (1.8mmol/L)
4. Very high or high cardiovascular risk
5. TG≤500 mg/dL(5.64 mmol/L)

Exclusion criteria:

1. Diagnosis of HoFH or HeFH
2. Uncontrolled hypertension
3. Uncontrolled hyperthyroidism or hypothyroidism
4. Severe renal dysfunction
5. Known sensitivity to any of the products to be administered during dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Mean percent change from baseline in low-density lipoprotein cholesterol (LDL-C) at week 48 | Week 48

SECONDARY OUTCOMES:
The percent of subjects with LDL-C reduction no less than 50% from baseline | Week 48
The percent of subjects with LDL-C<70mg/dL(1.8 mmol/L) | Week 48
The percent change in Lp(a),ApoB, non-HDL-c, ApoB/ApoA1 from baseline | Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China